CLINICAL TRIAL: NCT05717894
Title: Randomized, Post-marketing, Open-label, Observational, Non-interventional, Comparative, Controlled, Monocenter Study of the Efficacy and Safety of Mastodinone in Patients With Fibrocystic Breast Disease
Brief Title: Possibilities of Phytomedicine in Monotherapy of Benign Breast Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nazgul Omarbayeva (Other)
Responsible Party: Sponsor-Investigator, Nazgul Omarbayeva, Principal Scientist, Kazakh Institute of Oncology and Radiology
Organization: Kazakh Institute of Oncology and Radiology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MastoVit150
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Fibrocystic Breast Disease
MeSH Terms: conditions — Fibrocystic Breast Disease | interventions — Vitex agnus castus extract

STUDY DESIGN:
Intervention Model Description: all patients were randomized one-to-one into either the control group (n=72) or the treatment (primary) group (n=78) according to the order of admission to the hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment ( primary ) (Experimental)
  Interventions: Drug: Vitex Agnus Castus Extract
- Control (No Intervention)

INTERVENTIONS:
Drug: Vitex Agnus Castus Extract — The patient group received two pills containing 200mg of VAC daily for six months
  Other Names: Mastodynone
  Arms: Treatment ( primary )

SUMMARY:
The aim of this study is to evaluate the effectiveness of the use of the drug, containing Vitex agnus castus extract (VAC), in patients with fibrocystic breast disease . One hundred fifty women over 40 years old were randomized into patient (n=78) and control (n=72) groups. The groups were similar regarding age, nulliparity, menopause and abortion status, family history of breast cancer, alcohol consumption, and smoking. The patient group received two pills containing 200mg of VAC daily for six months, and all participants were evaluated by using a Visual Analogue Scale and ultrasound examination at baseline, 12th and 24th weeks.

DETAILED DESCRIPTION:
One hundred fifty patients presented at the Kazakh Institute of Oncology and Radiology diagnosed with FBD between January 2020, and May 2022 were prospectively enrolled in this study. The diagnosis was established based on complaints, palpation, and ultrasound findings. The patients over 40 years were also routinely screened by mammography to avoid breast cancer before including the study. Then, all patients were randomized one-to-one into either the control group (n=72) or the treatment (primary) group (n=78) according to the order of admission to the hospital. The envelope method was used so that the doctor and radiologist who performed the examination and ultrasound of the patients did not know which arm the patients were in.

Persistent pain was identified as a pain that lasts more than 3 months despite medication or treatment . The treatment group received two pills containing 200mg of VAC daily for six months, while the investigators followed the control group during the same period. Treatment responses were assessed using some subjective like the intensity of breast pain (from no pain=10 to unbearable pain=10), breast tenderness, and objective measures like palpable lumps and ultrasonographic examination performed at baseline, 12th and 24th weeks after the treatment by the same equipment and investigator. For the evaluation of breast pain at baseline and follow-up, a visual analogue scale marked from "no pain" to "unbearable pain" was used. Patients were asked to choose pictures of faces ranging from smiling to pain-contorted, conveying their perception of pain severity . Pain intensity was assessed using a visual analogue scale (VAS) in scores. The state of breast tissue was evaluated according to ultrasound findings; progression (increase in size and/or the number of cysts or fibrosis), stabilization (no clinically significant changes), and regression (partial or complete clinical response).

All participants read and signed written informed consent. The study was conducted at the Kazakh Institute of Oncology and Radiology based on a protocol proposed by the research team and approved by the Local Ethics committee according to principles of the World Medical Association (WMA) the Declaration of Helsinki 08/19 from 30th of October 2019.

Statistical analysis To compare the subgroups in terms of numerical variables, the normality was assessed by the Kolmogorov-Smirnov normality test, and the homogeneity of group variances was assessed by the Levene test. Mann-Whitney U test was used to determine the difference in the groups with median (minimum-maximum values) as descriptive statistics due to the skewed nature of those variables. Frequencies and percentages were presented to describe the categorical variables. The association between the groups and categorical variables was assessed with univariate analysis by the Pearson Chi-square test or fisher exact test, and the Bonferroni method was used to compare subgroups; if there was no difference between the groups, it was shown with the same letter, and if there was a difference, it was shown with a different letter. The IBM SPSS Statistics (version 25.0 for Windows, Chicago, IL, USA) was used, and p<0.05 was considered signiﬁcant for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* Must be able to visit the investigators at the appointesssd time.

Exclusion Criteria:

* refused to sign informed consent
* pregnant and breastfeeding
* has severe chronic comorbid diseases (cancer, diabetes mellitus, systemic blood diseases, neuralgia, suffering from mental illness or legally incompetent, e.g.)
* participated in another clinical trial

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | every 3 months up to 6 months
  Commonly used pain measurement scale: the 11-point numeric rating scale, the visual analogue scale (VAS) from no pain to unbearable pain, and the five-point categorical verbal rating scale. VAS scores: from 0 to 10: 0 - no pain; 1-3 - mild pain; 4-6 - moderate pain; 7-9 - severe pain; and 10 - unbearable pain
Ultrasound | every 3 months up to 6 months
  Ultrasound was used to assess the size of cysts, lumps, ducts, fibroadenomas

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh Institute of Oncology and Radiology, Almaty, Almaty Region, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: by URL link
URL: https://docs.google.com/spreadsheets/d/1zaLMY-FdG044O5Ms0OeDcVg1E4WDrmZA/edit?usp=sharing&ouid=107299945880128634706&rtpof=true&sd=true